CLINICAL TRIAL: NCT03275324
Title: Use of Integrated Pulmonary Index to Predict Post-Operative Respiratory Adverse Events in High Risk Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 1037010
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled patients: Surgical patients meeting enrollment criteria
  Interventions: Device: Capnostream20p

INTERVENTIONS:
Device: Capnostream20p — Observational study of patients connected to the Capnostream20p monitor.

SUMMARY:
The Capnostream 20p monitor by Medtronic is FDA-cleared and consists of a monitor which measures real-time respiratory status based on respiratory rate, pulse rate, pulse oximetry (SpO2) and end tidal carbon dioxide (etCO2) with a disposable nasal canula.

The integrated pulmonary index (IPI) is an algorithm driven parameter derived from non-invasive etCO2, respiratory rate, pulse rate and SpO2. Fuzzy logic is used to produce a value from 1-10 with 4 and under requiring intervention and 8-10 representing the normal range.

The purpose of this observational study is to determine if the IPI is associated with complications in the immediate postoperative period.

The study will enroll approximately 600 patients at 2 centers. Clinicians will be blinded to the IPI therefore this device will not be used to guide care in any way.

ELIGIBILITY:
Inclusion Criteria:

18 years or older Planned to undergo general anesthesia for surgery

Exclusion Criteria:

Pregnant Inability to consent Mechanically ventilated prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Respiratory Event | Up to 2 hours
  Respiratory complications occurring after surgery